CLINICAL TRIAL: NCT03012919
Title: Evaluation of an Active Decision Support System for Hemodynamic Optimization During High Risk Vascular Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Arabella Fischer, MD, Dr., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1967/2014
Record Dates: First submitted 2016-12-30; First posted 2017-01-06 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Feasibility; Active Decision Support System; Goal Directed Therapy
Keywords: active decision support system; goal directed therapy; Lidco; vascular surgery; hemodynamic optimization
MeSH Terms: interventions — Clinical Protocols

ARMS (1):
- active decision support system (GDT protocol) (Other): The active decision support system in this study is a goal directed therapy (GDT) protocol where threshold hemodynamic values are defined when to give fluid, vasopressors and inotropes. Hemodynamic values are measured with the LiDCOrapid device, which uses pulse contour analysis to continuously monitor cardiac output and respiratory variations in stroke volume (SVV).
  Interventions: Other: active decision support system

INTERVENTIONS:
Other: active decision support system — The active decision support system in this study is a goal directed therapy (GDT) protocol where threshold hemodynamic values are defined when to give fluid, vasopressors and inotropes. Hemodynamic values are measured with the LiDCOrapid device, which uses pulse contour analysis to continuously monitor cardiac output and respiratory variations in stroke volume (SVV).
  Other Names: goal directed therapy (GDT) protocol

SUMMARY:
Rivers et al. laid the foundation for modern hemodynamic and fluid management by establishing goal directed therapy (GDT) for the treatment of sepsis using fluid and inotropic and vasoactive agents. There have been many subsequent protocols to improve outcome in the operating room or in the ICU. These are mainly passive decision support systems. Active clinical decision support systems using fluid and pharmacologic agents to improve intraoperative hemodynamics are not really found.

The investigators developed an active clinical decision support system based on an institutional GDT-protocol using fluid, vasopressors and inotropes using the LiDCOrapid device.

The goal of the study was to check the feasibility of an active clinical decision support system to optimize hemodynamics during high risk vascular surgery based on the principles of GDT implementing fluid, vasopressors and inotropes.

ELIGIBILITY:
Inclusion Criteria:

* elective major vascular surgery such as peripheral arterial surgery and open abdominal aortic surgery except for carotid artery surgery

Exclusion Criteria:

* patients under 18 years of age
* absence of cardiac sinus rhythm at induction of anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
number of interventions done according to the active decision support system (GDT protocol) | through study completion, an average of 6 months
  The number of interventions done according to the active decision support system (GDT protocol) is calculated.
duration of use of active decision support system | through study completion, an average of 6 months
  The absolute duration of use and relative duration of use (in relation to the duration of surgery) of the active decision support system are calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Dworschak, Prof. Dr., Study Director — Medical University of Vienna; Michael Hiesmayr, Prof. Dr., Study Director — Medical University of Vienna; Johannes Menger, Dr., Principal Investigator — Medical University of Vienna; Arabella Fischer, Dr., Principal Investigator — Medical University of Vienna

REFERENCES:
- [Background] Fitzgerald M, Cameron P, Mackenzie C, Farrow N, Scicluna P, Gocentas R, Bystrzycki A, Lee G, O'Reilly G, Andrianopoulos N, Dziukas L, Cooper DJ, Silvers A, Mori A, Murray A, Smith S, Xiao Y, Stub D, McDermott FT, Rosenfeld JV. Trauma resuscitation errors and computer-assisted decision support. Arch Surg. 2011 Feb;146(2):218-25. doi: 10.1001/archsurg.2010.333. PMID 21339436
- [Background] Feldheiser A, Conroy P, Bonomo T, Cox B, Garces TR, Spies C; Anaesthesia Working Group of the Enhanced Recovery After Surgery (ERAS(R)) Society; Enhanced Recovery After Surgery Society. Development and feasibility study of an algorithm for intraoperative goaldirected haemodynamic management in noncardiac surgery. J Int Med Res. 2012;40(4):1227-41. doi: 10.1177/147323001204000402. PMID 22971475
- [Background] Sondergaard S, Wall P, Cocks K, Parkin WG, Leaning MS. High concordance between expert anaesthetists' actions and advice of decision support system in achieving oxygen delivery targets in high-risk surgery patients. Br J Anaesth. 2012 Jun;108(6):966-72. doi: 10.1093/bja/aes037. Epub 2012 Mar 16. PMID 22427342
- [Background] Sahota N, Lloyd R, Ramakrishna A, Mackay JA, Prorok JC, Weise-Kelly L, Navarro T, Wilczynski NL, Haynes RB; CCDSS Systematic Review Team. Computerized clinical decision support systems for acute care management: a decision-maker-researcher partnership systematic review of effects on process of care and patient outcomes. Implement Sci. 2011 Aug 3;6:91. doi: 10.1186/1748-5908-6-91. PMID 21824385